CLINICAL TRIAL: NCT04764110
Title: Short-term Impact of Cyplexinol® on Inflammatory Status and Related Measures in Men and Women With Self-reported Joint Pain
Brief Title: Short-term Impact of Cyplexinol® on Self-reported Joint Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Memphis (Other)
Collaborators: ZyCal Bioceuticals (Unknown)
Responsible Party: Principal Investigator, Richard Bloomer, Dean of the College of Health Sciences, University of Memphis
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: PRO-FY2021-6
Record Dates: First submitted 2021-02-18; First posted 2021-02-21 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Joint Pain
Keywords: Cyplexinol; Inflammation
MeSH Terms: conditions — Arthralgia; Inflammation

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized, control
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cyplexinol (Experimental): 900 mg daily (2 capsules) for 15 days
  Interventions: Dietary Supplement: Cyplexinol
- Placebo (Placebo Comparator): 2 capsules daily for 15 days
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Cyplexinol — partially hydrolyzed Collagen and its associated proteins including Bone Morphogenetic Proteins (BMPs)
  Arms: Cyplexinol
Other: Placebo — Maltodextrin
  Arms: Placebo

SUMMARY:
In this study, the impact of 900 mg Cyplexinol® taken daily on joint pain over a period of 15 days in comparison with a placebo will be determined using a cross-over double blind design with a 13 day wash out period. In addition, we will measure cytokine production and related variables during the two hour after subjects ingest a single dosage of Cyplexinol® or placebo on days 1 and 15.

DETAILED DESCRIPTION:
Chronic inflammation can induce joint pain, which is a common problem among adult men and women. ZyCal Bioceuticals is a manufacturer of natural ingredients and finished nutritional supplements to support bone and joint health in humans. The core ingredient in all ZyCal products is Cyplexinol® (a Bone Morphogenetic Protein [BMP] Complex). BMP complexes have been shown to activate mesenchymal stem cells to help the body regenerate osteoblasts and chondrocytes. BMPs were initially identified in the 1970's as osteogenic factors which stimulate activation, proliferation, and differentiation of osteoprogenitor cells by binding BMP receptors and subsequent signaling through the SMAD pathway. BMPs have also been shown to reduce inflammation and promote healthy inflammatory signaling in joints and other tissues.

Cyplexinol® is delivered in the dietary supplement called Ostinol™, which has been safely used in oral form by thousands of people since 2007 for bone and joint health. Currently Cyplexinol® is considered a dietary supplement ingredient and has been awarded GRAS (generally recognized as safe).

Studies have been conducted to evaluate the safety and efficacy of Cyplexinol® as a dietary supplement for joint health (Garian, 2012; Scaffidi, 2017). Dosages of 150mg Cyplexinol® have been compared to a placebo (negative control) alone or in combination with glucosamine /chondroitin in randomized controlled trials for 4 -12 weeks. Endpoints examined have included joint stiffness, inflammation, pain, and overall quality of life. However, to date, no short-term studies have been conducted using Cyplexinol®, nor have any acute studies evaluated the impact of this agent on immune function.

In this study, the impact of 900 mg Cyplexinol® taken daily on joint pain over a period of 15 days in comparison with a placebo will be determined using a cross-over double blind design with a 13 day wash out period. In addition, we will measure cytokine production and related variables during the two hour post ingestion period after subjects ingest a single dosage of Cyplexinol® or placebo on days 1 and 15.

ELIGIBILITY:
Inclusion Criteria:

* body mass index (BMI) between 18-29.9 kg/m2 (not obese)
* no consumption of alcohol-containing beverages within 48 hours of testing
* experiencing self-reported joint pain with a minimum pain rating of 3/10 for at least the past 30 days
* engaged in structured exercise 2 or more days per week for the past 6 months or longer
* a negative verbal pre-study drug screen (alcohol abuse, amphetamines, benzodiazepines, cocaine, opioids, phencyclidine, barbiturates, cotinine), no history of use of illicit drugs or other substances of abuse within 12 months of the screening visit

Exclusion Criteria:

* pregnant
* tobacco user
* active infection or illness of any kind
* rheumatic or osteoarthritic diagnosis
* Using anti-inflammatory medicines, pain medications, or dietary supplements (or not willing to cease for one-month prior to participation and throughout study)

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-03-17 (Actual); Primary Completion 2022-01-28 (Actual); Study Completion 2022-01-28 (Actual)

PRIMARY OUTCOMES:
TNF-alpha | baseline of day 1
  TNF-alpha measured in blood
TNF-alpha | baseline of day 15
  TNF-alpha measured in blood
TNF-alpha | 60 min after treatment ingestion of day 1
  TNF-alpha measured in blood
TNF-alpha | 60 min after treatment ingestion of day 15
  TNF-alpha measured in blood
TNF-alpha | 120 min after treatment ingestion of day 1
  TNF-alpha measured in blood
TNF-alpha | 120 min after treatment ingestion of day 15
  TNF-alpha measured in blood
IL-6 | baseline of day 1
  IL-6 measured in blood
IL-6 | baseline of day 15
  IL-6 measured in blood
IL-6 | 60 min after treatment ingestion of day 1
  IL-6 measured in blood
IL-6 | 60 min after treatment ingestion of day 15
  IL-6 measured in blood
IL-6 | 120 min after treatment ingestion of day 1
  IL-6 measured in blood
IL-6 | 120 min after treatment ingestion of day 15
  IL-6 measured in blood
IL-10 | baseline of day 1
  IL-10 measured in blood
IL-10 | baseline of day 15
  IL-10 measured in blood
IL-10 | 60 min after treatment ingestion of day 1
  IL-10 measured in blood
IL-10 | 60 min after treatment ingestion of day 15
  IL-10 measured in blood
IL-10 | 120 min after treatment ingestion of day 1
  IL-10 measured in blood
IL-10 | 120 min after treatment ingestion of day 15
  IL-10 measured in blood
IL-1beta | baseline of day 1
  IL-1beta measured in blood
IL-1beta | baseline of day 15
  IL-1beta measured in blood
IL-1beta | 60 min after treatment ingestion of day 1
  IL-1beta measured in blood
IL-1beta | 60 min after treatment ingestion of day 15
  IL-1beta measured in blood
IL-1beta | 120 min after treatment ingestion of day 1
  IL-1beta measured in blood
IL-1beta | 120 min after treatment ingestion of day 15
  IL-1beta measured in blood
osteocalcin | baseline day 1
  osteocalcin measured in blood
osteocalcin | baseline day 15
  osteocalcin measured in blood
osteocalcin | 60 min after treatment ingestion of day 1
  osteocalcin measured in blood
osteocalcin | 60 min after treatment ingestion of day 15
  osteocalcin measured in blood
osteocalcin | 120 min after treatment ingestion of day 1
  osteocalcin measured in blood
osteocalcin | 120 min after treatment ingestion of day 15
  osteocalcin measured in blood
alkaline phosphatase | baseline day 1
  alkaline phosphatase measured in blood
alkaline phosphatase | baseline day 15
  alkaline phosphatase measured in blood
alkaline phosphatase | 60 min after treatment ingestion of day 1
  alkaline phosphatase measured in blood
alkaline phosphatase | 60 min after treatment ingestion of day 15
  alkaline phosphatase measured in blood
alkaline phosphatase | 120 min after treatment ingestion of day 1
  alkaline phosphatase measured in blood
alkaline phosphatase | 120 min after treatment ingestion of day 15
  alkaline phosphatase measured in blood
Bone Morphogenetic Protein | baseline day 1
  Bone Morphogenetic Protein measured in blood
Bone Morphogenetic Protein | baseline day 15
  Bone Morphogenetic Protein measured in blood
Bone Morphogenetic Protein | 60 min after treatment ingestion of day 1
  Bone Morphogenetic Protein measured in blood
Bone Morphogenetic Protein | 60 min after treatment ingestion of day 15
  Bone Morphogenetic Protein measured in blood
Bone Morphogenetic Protein | 120 min after treatment ingestion of day 1
  Bone Morphogenetic Protein measured in blood
Bone Morphogenetic Protein | 120 min after treatment ingestion of day 15
  Bone Morphogenetic Protein measured in blood
Joint pain visual analog scale | Day 1 of treatment
  A 100mm visual analog scale will be used to assess joint pain. Scores range from 0 (subject strongly disagreeing with prompt) to 100 (strongly agree).
Joint pain visual analog scale | Day 15 of treatment
  A 100mm visual analog scale will be used to assess joint pain. Scores range from 0 (subject strongly disagreeing with prompt) to 100 (strongly agree).
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Day 1 of treatment
  The WOMAC measures five items for pain (score range 0-20), two for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68) with 0 being none and high values being most.
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Day 15 of treatment
  The WOMAC measures five items for pain (score range 0-20), two for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68) with 0 being none and high values being most.

SECONDARY OUTCOMES:
Dietary intake | Day 1 of treatment
  Dietary intake of subjects for 3-days prior to testing days analyzed using Food Processor Pro software for total calories, macro- and micro-nutrient composition
Dietary intake | Day 15 of treatment
  Dietary intake of subjects for 3-days prior to testing days analyzed using Food Processor Pro software for total calories, macro- and micro-nutrient composition

CONTACTS AND LOCATIONS:
Overall Officials: Richard Bloomer, PhD, Principal Investigator — University of Memphis
Locations (1):
- Center for Nutraceutical and Dietary Supplement Reseach, Memphis, Tennessee, United States